CLINICAL TRIAL: NCT03102034
Title: Phase I Placebo-Controlled Study of the Infectivity, Safety and Immunogenicity of a Single Dose of a Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine, D46/NS2/N/ΔM2-2-HindIII, Lot RSV#011B, Delivered as Nose Drops to RSV-Seronegative Infants 6 to 24 Months of Age
Brief Title: Evaluating the Infectivity, Safety, and Immunogenicity of a Single Dose of a Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine (D46/NS2/N/ΔM2-2-HindIII) in RSV-Seronegative Infants 6 to 24 Months of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMPAACT 2013; 30074 (Registry Identifier: DAIDS-ES Registry Number); NCT03099291 (obsolete NCT alias)
Record Dates: First submitted 2017-03-23; First posted 2017-04-05 (Actual); Results first posted 2019-06-14 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RSV D46/NS2/N/ΔM2-2-HindIII Vaccine (Experimental): Participants received a single dose of the D46/NS2/N/ΔM2-2-HindIII vaccine at study entry (Day 0).
  Interventions: Biological: D46/NS2/N/ΔM2-2-HindIII
- Placebo (Placebo Comparator): Participants received a single dose of placebo at study entry (Day 0).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: D46/NS2/N/ΔM2-2-HindIII — 10^5 plaque-forming units (PFU) per 0.5ml vaccine; administered as nose drops
  Arms: RSV D46/NS2/N/ΔM2-2-HindIII Vaccine
Biological: Placebo — Isotonic diluent; administered as nose drops
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety, infectivity, and immunogenicity of a single dose of a recombinant live-attenuated respiratory syncytial virus (RSV) vaccine in RSV-seronegative infants and children 6 to 24 months of age.

This study was a companion study to CIR 313.

DETAILED DESCRIPTION:
Human respiratory syncytial virus (RSV) is the most common viral cause of serious acute lower respiratory illness (LRI) in infants and children under 5 years of age worldwide. This study evaluated the safety, infectivity, and immunogenicity of a single dose of RSV D46/NS2/N/ΔM2-2-HindIII, a recombinant live-attenuated RSV vaccine, in RSV-seronegative infants and children 6 to 24 months of age.

Participants were randomly assigned to receive a single dose of the D46/NS2/N/ΔM2-2-HindIII vaccine or placebo (administered as nose drops) at study entry (Day 0).

Participants could be enrolled in the study outside of RSV season (between April 1 and October 14 for most sites or-for sites with local RSV seasons that start earlier-as specified on a site-by-site basis in the Manual Of Procedures). All participants remained on study until they completed the post-RSV season visit between April 1 and April 30 in the calendar year following enrollment. Participants' total study duration was between 6 and 13 months, depending on when they enrolled in the study. Participants attended several study visits throughout the study, which included physical examinations, blood collection, and nasal washes. Participants' parents or guardians were contacted by study staff at various times during the study to monitor participants' health.

ELIGIBILITY:
Inclusion Criteria:

* Good health based on review of the medical record, history, and physical examination, without evidence of chronic disease.
* Parents/guardians willing and able to provide written informed consent as described in the protocol.
* Seronegative for RSV antibody, defined as a serum RSV-neutralizing antibody titer less than 1:40 at screening from a sample collected no more than 42 days prior to inoculation. Note: results from specimens collected during screening for any study of an RSV vaccine developed by the Laboratory of Infectious Diseases (LID) (NIAID, NIH) were acceptable as long as within the 42-day window.
* Growing at a normal velocity for age (as demonstrated on a standard growth chart) AND

  * If less than 1 year of age: current height and weight above the 5th percentile
  * If 1 year of age or older: current height and weight above the 3rd percentile for age.
* Received routine immunizations appropriate for age (as per national Center for Disease Control Advisory Committee on Immunization Practices [ACIP]). Note: if rotavirus immunization was delayed, "catch-up" rotavirus immunization was indicated only if the participant was age-eligible per ACIP.
* Expected to be available for the duration of the study.
* If born to an HIV-infected woman, participant must not have been breastfed and must have had documentation of 2 negative HIV nucleic acid (RNA or DNA) test results from samples collected on different dates with both collected when greater than or equal to 4 weeks of age and at least one collected when greater than or equal to 16 weeks of age, and no positive HIV nucleic acid (RNA or DNA) test; or 2 negative HIV antibody tests, both from samples collected at greater than or equal to 24 weeks of age.

Exclusion Criteria:

* Known or suspected HIV infection or impairment of immunological functions.
* Receipt of immunosuppressive therapy, including any systemic, including either nasal or inhaled, corticosteroids within 28 days of enrollment. Note: Cutaneous (topical) steroid treatment was not an exclusion.
* Bone marrow/solid organ transplant recipient.
* Major congenital malformations (such as congenital cleft palate) or cytogenetic abnormalities.
* Previous receipt of a licensed or investigational RSV vaccine (or placebo in any IMPAACT RSV study) or previous receipt of or planned administration of any anti-RSV product (such as ribavirin or RSV immunoglobulin [IG] or RSV monoclonal antibody [mAb]).
* Previous anaphylactic reaction.
* Previous vaccine-associated adverse reaction that was Grade 3 or above.
* Known hypersensitivity to any study product component.
* Heart disease. Note: Participants with cardiac abnormalities documented to be clinically insignificant and requiring no treatment may be enrolled.
* Lung disease, including any history of reactive airway disease or medically diagnosed wheezing.
* Member of a household that contained, or would contain, an infant who was less than 6 months of age at the enrollment date through Day 28.
* Member of a household that contains another child who was, or was scheduled to be, enrolled in IMPAACT 2011, 2012 or 2013 or another study evaluating an intranasal live-attenuated RSV vaccine, AND there had been or would be an overlap in residency during that other child's participation in the study's Acute Phase (Days 0 to 28).
* Member of a household that contained an immunocompromised individual, including, but not limited to:

  * a person who was greater than or equal to 6 years of age with HIV-related immunodeficiency, defined as having a most recent CD4 T lymphocyte cell count less than 300 cells/mm^3. CD4 T lymphocyte count must have been measured within 6 months prior to enrollment, or
  * a person age 1 year up to less than 6 years with HIV-related immunodeficiency, defined as having a most recent CD4 T lymphocyte cell percentage less than 25 or CD4 T lymphocyte count less than 750 cells/mm^3 (if both values are available, use the lower of the two). CD4 T lymphocyte parameter must have been measured within the 6 months prior to enrollment; or
  * a person age less than 1 year with HIV-related immunodeficiency, defined as having a most recent CD4 T lymphocyte cell percentage less than 30 or CD4 T lymphocyte count less than 1000 cells/mm^3 (if both values are available, use the lower of the two). CD4 T lymphocyte parameter must have been measured within the 6 months prior to enrollment; or
  * a person who had received chemotherapy within the 12 months prior to enrollment; or
  * a person receiving immunosuppressant agents; or
  * a person living with a solid organ or bone marrow transplant.

Verbal report of CD4 T cell lymphocyte was sufficient documentation if the parent/guardian was confident of history.

* Attended a daycare facility and shared a room with infants less than 6 months of age, and parent/guardian was unable or unwilling to suspend daycare for 28 days following inoculation.
* Any of the following events at the time of enrollment:

  * fever (rectal temperature of greater than or equal to 100.4°F (38°C)), or
  * upper respiratory signs or symptoms (rhinorrhea, cough, or pharyngitis) or
  * nasal congestion significant enough to interfere with successful inoculation, or
  * otitis media.
* Receipt of the following prior to enrollment:

  * any inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior
* Scheduled administration of the following after planned inoculation:

  * inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days after, or
  * any live vaccine other than rotavirus in the 28 days after, or
  * another investigational vaccine or investigational drug in the 56 days after
* Receipt of immunoglobulin, any antibody products, or any blood products within the past 6 months
* Receipt of any of the following medications within 3 days of study enrollment:

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medication except as listed below

Permitted concomitant medications (prescription or non-prescription) include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) cutaneous (topical) steroids, topical antibiotics, and topical antifungal agents.

* Receipt of salicylate (aspirin) or salicylate-containing products within the 28 days prior to enrollment.
* Born at less than 34 weeks gestation.
* Born at less than 37 weeks gestation and less than 1 year of age at the time of enrollment.
* Suspected or documented developmental disorder, delay, or other developmental problem.
* Previous receipt of supplemental oxygen therapy in a home setting.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth (Betsy) J. McFarland, MD, Study Chair — University of Colorado School of Medicine and Children's Hospital Colorado, Pediatric Infectious Diseases
Locations (10):
- United States (10):
  - Usc La Nichd Crs, Los Angeles, California
  - David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Emory University School of Medicine NICHD CRS, Atlanta, Georgia
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Johns Hopkins University Center for Immunization Research, Baltimore, Maryland
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee

REFERENCES:
- [Derived] McFarland EJ, Karron RA, Muresan P, Cunningham CK, Perlowski C, Libous J, Oliva J, Jean-Philippe P, Moye J, Schappell E, Barr E, Rexroad V, Fearn L, Cielo M, Wiznia A, Deville JG, Yang L, Luongo C, Collins PL, Buchholz UJ. Live-Attenuated Respiratory Syncytial Virus Vaccine With M2-2 Deletion and With Small Hydrophobic Noncoding Region Is Highly Immunogenic in Children. J Infect Dis. 2020 Jun 11;221(12):2050-2059. doi: 10.1093/infdis/jiaa049. PMID 32006006
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.0, November 2014 — http://rsc.tech-res.com/docs/default-source/safety/daids_ae_grading_table_v2_nov2014.pdf
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.tech-res.com/docs/default-source/safety/manual_for_expedited_reporting_aes_to_daids_v2.pdf?sfvrsn=12

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from April to October 2017. Participants were recruited from medical clinics.
Period: Overall Study
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo
Started | 21 | 11
Completed | 20 | 11
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was participants who received inoculation.
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo | Total
Number analyzed (Participants) | 21 | 11 | 32
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 9 [7 to 13] | 9 [6 to 15] | 9 [7 to 13.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 6 | 18
  Not Hispanic or Latino | 9 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 14 | 6 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 21 | 11 | 32
Serum RSV-neutralizing antibody titers [Median (Inter-Quartile Range); unit: log 2 titers] — Data values are presented as log 2 titers.
  log 2 titers | 2.3 [2.3 to 2.3] | 2.3 [2.3 to 3.3] | 2.3 [2.3 to 3.3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events (AEs) by Grade
Description: Solicited adverse events included fever; otitis media; upper respiratory illness (URI); lower respiratory illness (LRI) and cough (without LRI). The number of participants who experienced solicited adverse events was presented. A participant was only counted once in each solicited AE category, and that was in the line corresponding to the highest grade adverse event they had in that category. These events were graded (Grade 1-mild to Grade 4-life-threatening) following protocol-defined grading system outlined in Table 3 and Table 4 in the protocol document.
Time Frame: Measured from Day 0 through Day 28
Population: Study participants who received inoculation were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo
Number analyzed (Participants) | 21 | 11
Participants
  Fever: Did not have this AE | 17 | 9
  Fever: Grade 1 | 3 | 1
  Fever: Grade 2 | 1 | 1
  Fever: Grade 3 | 0 | 0
  Fever: Grade 4 | 0 | 0
  Otitis Media: Did not have this AE | 21 | 11
  Otitis Media: Grade 1 | 0 | 0
  Otitis Media: Grade 2 | 0 | 0
  Otitis Media: Grade 3 | 0 | 0
  Otitis Media: Grade 4 | 0 | 0
  Upper Respiratory Illness (URI): Did not have this AE | 6 | 10
  Upper Respiratory Illness (URI): Grade 1 | 15 | 1
  Upper Respiratory Illness (URI): Grade 2 | 0 | 0
  Upper Respiratory Illness (URI): Grade 3 | 0 | 0
  Upper Respiratory Illness (URI): Grade 4 | 0 | 0
  Lower Respiratory Illness (LRI): Did not have this AE | 21 | 11
  Lower Respiratory Illness (LRI): Grade 1 | 0 | 0
  Lower Respiratory Illness (LRI): Grade 2 | 0 | 0
  Lower Respiratory Illness (LRI): Grade 3 | 0 | 0
  Lower Respiratory Illness (LRI): Grade 4 | 0 | 0
  Cough, without LRI: Did not have this AE | 9 | 11
  Cough, without LRI: Grade 1 | 12 | 0
  Cough, without LRI: Grade 2 | 0 | 0
  Cough, without LRI: Grade 3 | 0 | 0
  Cough, without LRI: Grade 4 | 0 | 0
Statistical Analysis 1: Comparison: RSV D46/NS2/N/ΔM2-2-HindIII Vaccine; Test type: Other; % vaccine recipients with solicited AEs = 76, 90% CI 2-sided [56 to 90] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 2: Comparison: Placebo; Test type: Other; % placebo recipients with solicited AEs = 18, 90% CI 2-sided [3 to 47] — Confidence intervals were Exact Clopper-Pearson

2. Primary Outcome: Number of Participants With Unsolicited AEs by Grade
Description: Unsolicited adverse events were other events, not included in the solicited AEs. The number of participants who experienced solicited adverse events was presented. A participant was only counted once in each unsolicited AE category, and that was in the line corresponding to the highest grade adverse event they had in that category. AE grading (Grade 1- mild to Grade 4-life-threatening) was done by DAIDS AE Grading table v2.0 (see References).
Time Frame: Measured from Day 0 through Day 28
Population: Study participants who received inoculation were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo
Number analyzed (Participants) | 21 | 11
Participants
  Diarrhea, vomiting: Did not have this AE | 17 | 11
  Diarrhea, vomiting: Grade 1 | 4 | 0
  Diarrhea, vomiting: Grade 2 | 0 | 0
  Diarrhea, vomiting: Grade 3 | 0 | 0
  Diarrhea, vomiting: Grade 4 | 0 | 0
  Epistaxis: Did not have this AE | 20 | 10
  Epistaxis: Grade 1 | 1 | 1
  Epistaxis: Grade 2 | 0 | 0
  Epistaxis: Grade 3 | 0 | 0
  Epistaxis: Grade 4 | 0 | 0
  Nasal congestion: Did not have this AE | 20 | 11
  Nasal congestion: Grade 1 | 1 | 0
  Nasal congestion: Grade 2 | 0 | 0
  Nasal congestion: Grade 3 | 0 | 0
  Nasal congestion: Grade 4 | 0 | 0
  Sneezing: Did not have this AE | 20 | 11
  Sneezing: Grade 1 | 1 | 0
  Sneezing: Grade 2 | 0 | 0
  Sneezing: Grade 3 | 0 | 0
  Sneezing: Grade 4 | 0 | 0
  Eczema, Diaper rash: Did not have this AE | 19 | 11
  Eczema, Diaper rash: Grade 1 | 2 | 0
  Eczema, Diaper rash: Grade 2 | 0 | 0
  Eczema, Diaper rash: Grade 3 | 0 | 0
  Eczema, Diaper rash: Grade 4 | 0 | 0
  Middle ear effusion: Did not have this AE | 20 | 11
  Middle ear effusion: Grade 1 | 1 | 0
  Middle ear effusion: Grade 2 | 0 | 0
  Middle ear effusion: Grade 3 | 0 | 0
  Middle ear effusion: Grade 4 | 0 | 0
  Irritability: Did not have this AE | 20 | 11
  Irritability: Grade 1 | 1 | 0
  Irritability: Grade 2 | 0 | 0
  Irritability: Grade 3 | 0 | 0
  Irritability: Grade 4 | 0 | 0
  Lymphadenopathy: Did not have this AE | 20 | 11
  Lymphadenopathy: Grade 1 | 1 | 0
  Lymphadenopathy: Grade 2 | 0 | 0
  Lymphadenopathy: Grade 3 | 0 | 0
  Lymphadenopathy: Grade 4 | 0 | 0
Statistical Analysis 1: Comparison: RSV D46/NS2/N/ΔM2-2-HindIII Vaccine; Test type: Other; % vaccinees with unsolicited AEs = 24, 90% CI 2-sided [10 to 44] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 2: Comparison: Placebo; Test type: Other; % placebo with unsolicited AEs = 9, 90% CI 2-sided [0 to 36] — Confidence intervals were Exact Clopper-Pearson

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) was an AE, whether considered related to the study product or not, that:
  * Resulted in death during the period of protocol-defined surveillance
  * Was life threatening: defined as an event in which the patient was at immediate risk of death at the time of the event; it did not refer to an event that hypothetically might have caused death were it more severe
  * Required inpatient hospitalization (or prolongation of existing hospitalization): defined as at least an overnight stay in the hospital or emergency ward for treatment that would have been inappropriate if administered in the outpatient setting
  * Resulted in a persistent or significant disability/incapacity
  * Was a congenital anomaly or birth defect
  * Was an important medical event that might not be immediately life threatening or result in death or hospitalization but might jeopardize the patient or might require intervention to prevent one of the outcomes listed above.
Time Frame: Measured from Day 0 through Day 56
Population: Study participants who received inoculation were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo
Number analyzed (Participants) | 21 | 11
Participants | 0 | 0

4. Primary Outcome: Number of Participants Infected With RSV Vaccine Virus
Description: Defined as 1) vaccine virus identified in a nasal wash from Study Day 0-28 (a binary outcome based on nasal washes) and/or 2) greater than or equal to 4-fold rise in RSV-neutralizing antibody titer from Study Day 0 and 56.
Time Frame: Measured at Days 0, 3, 5, 7, 10, 12, 14, 17, and 28 for nasal washes, and at Days 0, 56 for serum RSV-neutralizing antibodies
Population: Study participants who received inoculation were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo
Number analyzed (Participants) | 21 | 11
Participants | 21 | 0

5. Primary Outcome: Peak Titer of Vaccine Virus Shed
Description: This is the highest value per participant of the titer of vaccine virus shed. It was measured by culture. Only participants who met the definition of infection with vaccine virus were included.
Time Frame: Measured at Days 0, 3, 5, 7, 10, 12, 14, 17, and 28
Population: Only participants who met the definition of infection with vaccine virus were included.
Measure: Median (Inter-Quartile Range); unit: log10 PFU/mL
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo
Number analyzed (Participants) | 21 | 0
log10 PFU/mL | 3.5 [2.9 to 3.8] |

6. Primary Outcome: Duration of Vaccine Virus Shedding in Nasal Washes
Description: Determined separately by a) culture and b) reverse transcription polymerase chain reaction (RT-PCR)
Time Frame: Measured at Days 0, 3, 5, 7, 10, 12, 14, 17, and 28. Last day positive is reported.
Population: Only participants who met the definition of infection with vaccine virus were included.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo
Number analyzed (Participants) | 21 | 0
days
  Culture positive | 10 [7 to 12] |
  RT-PCR positive | 14 [12 to 17] |

7. Primary Outcome: Number of Participants With a Greater Than or Equal to 4-fold Rise in Serum RSV-neutralizing Antibody Titer
Description: Immunogenicity was assessed pre-inoculation, and at approximately 2 months post-inoculation (Study Day 56). Antibody responses were defined as a greater than or equal to 4-fold increase in titer in paired specimens, between pre-inoculation and post-inoculation time points.
Time Frame: Measured at Day 0 and Day 56
Population: Study participants who received inoculation were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo
Number analyzed (Participants) | 21 | 11
Participants | 20 | 0
Statistical Analysis 1: Comparison: RSV D46/NS2/N/ΔM2-2-HindIII Vaccine vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — Due to unequal sample sizes, a 1-sided Fisher's exact test was used to test the hypothesis that proportions of greater than or equal to 4-fold rises were higher in the vaccinated than in the placebo group. Statistical significance level was 0.05

8. Primary Outcome: Serum Antibody Responses to RSV F Glycoprotein as Assessed by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Immunogenicity was assessed at approximately 2 months post-inoculation (Study Day 56).
Time Frame: Measured at Day 56
Population: Study participants who received inoculation were included.
Measure: Median (Inter-Quartile Range); unit: log 2 titers
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo
Number analyzed (Participants) | 21 | 11
log 2 titers | 15.7 [13.9 to 15.7] | 8.1 [6 to 9.1]
Statistical Analysis 1: Comparison: RSV D46/NS2/N/ΔM2-2-HindIII Vaccine vs Placebo; Test type: Superiority; p < 0.001, Log Rank — The threshold for statistical significance is 0.05

9. Secondary Outcome: Number of Participants Who Had Symptomatic, Medically Attended Respiratory and Febrile Illness, Among Those Who Experienced Natural Infection With wt RSV During the Subsequent RSV Season
Description: The number of participants who had RSV-associated, medically attended, acute respiratory illness (RSV-MAARI) or RSV-associated, medically attended, acute lower respiratory illness (RSV-MAALRI) among those who had RSV detected in nasal washes or greater than or equal to 4 fold rise in serum antibodies during the subsequent RSV season were presented.
Time Frame: Measured from November 1st through participant's post-RSV season surveillance visit
Population: Only participants who had RSV detected in nasal washes or greater than or equal to 4 fold rise in serum antibodies during the subsequent RSV season were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo
Number analyzed (Participants) | 6 | 4
Participants
  RSV-MAARI | 2 | 3
  RSV-MAALRI | 0 | 1

10. Secondary Outcome: Magnitude of Serum RSV-neutralizing Antibody Responses in the Vaccine and Placebo Recipients Who Experienced Natural Infection With wt RSV During the Subsequent RSV Season.
Description: Only participants who had RSV detected in nasal washes or a greater than or equal to 4-fold rise in serum antibodies during the subsequent RSV season were included. RSV-neutralizing antibody titers were measured pre- and post-RSV surveillance season.
Time Frame: Measured through participant's last study visit, up to a total of 6 to 13 months depending on when participants enrolled in the study
Population: Only participants who had RSV detected in nasal washes or a greater than or equal to 4-fold rise in serum antibodies during the subsequent RSV season were included.
Measure: Median (Inter-Quartile Range); unit: log 2 titers
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo
Number analyzed (Participants) | 6 | 4
log 2 titers
  Pre-RSV surveillance | 6.3 [4.5 to 7.7] | 2.3 [2.3 to 2.8]
  Post-RSV Surveillance | 10.4 [6.4 to 11.0] | 7.1 [5.9 to 8.8]

11. Secondary Outcome: Number of Participants With B Cell Responses to Vaccine
Description: A B cell response to vaccine is indicated by a greater than or equal to 4-fold change in serum antibody titers to RSV F glycoprotein between the pre- and post-inoculation time points.
Time Frame: Measured at day 0 and Day 56
Population: All participants who received inoculation were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV D46/NS2/N/ΔM2-2-HindIII Vaccine | Placebo
Number analyzed (Participants) | 21 | 11
Participants | 21 | 0

12. Other Pre Specified Outcome: Frequency of Mucosal Antibody Responses to Vaccine
Description: Determined from nasal wash samples. This outcome has been changed from a secondary outcome measure to an 'other pre-specified' outcome measure. Since this outcome measure relies on previously untested assays to reliably quantify RSV specific mucosal antibodies from nasal wash samples, it was changed to other pre-specified to fit with its intended analysis type.
Time Frame: Measured at Day 0, 28 and 56
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From study entry to end of study. The duration of follow-up for a given participant was between 6 and 13 months depending on time of enrollment.
Description: From day 0-28, all SAEs, solicited AEs, and unsolicited AEs, with the exception of the following if not treated with prescription medication or over the counter medications with antipyretic properties: diaper rashes, teething pain, and spitting up. SAEs and LRIs were reported according to DAIDS EAE Manual V2.0 (see References).
  From day 29-56, SAEs were collected. After day 56, from November 1 - March 31 of the following year, medically attended fever, LRI, URI and otitis media were collected.
Groups:
- Vaccine: Participants received a single dose of the D46/NS2/N/ΔM2-2-HindIII vaccine at study entry (Day 0).
  D46/NS2/N/ΔM2-2-HindIII: 10^5 plaque-forming units (PFU) per 0.5ml vaccine; administered as nose drops
- Placebo: Participants received a single dose of placebo study entry (Day 0). Placebo: Isotonic diluent, administered as nose drops
Arm/Group | Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/11
Other Adverse Events (participants affected / at risk) | 17/21 | 10/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=21) | Placebo (N=11)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 0
Infantile vomiting (Gastrointestinal disorders) | 2 | 0
Pyrexia (General disorders) | 10 | 6
Conjunctivitis viral (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 5 | 2
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT03102034/Prot_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan, Version 1.0 (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT03102034/SAP_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan, Version 3.1 (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT03102034/SAP_003.pdf